CLINICAL TRIAL: NCT07156539
Title: A Study of HS-20094 Versus Dulaglutide Once Weekly as Add-on Therapy to Metformin Monotherapy or in Combination With SGLT2 Inhibitors in Participants With Type 2 Diabete
Brief Title: A Phase 3 Study of HS-20094 in Patients With T2DM
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-20094-303
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group A (Experimental): HS-20094-low dose
  Interventions: Drug: HS-20094 Injection
- Treatment Group B (Experimental): HS-20094-high dose
  Interventions: Drug: HS-20094 Injection
- Treatment Group C (Active Comparator): Dulaglutide -1.5mg
  Interventions: Drug: Dulaglutide Injection

INTERVENTIONS:
Drug: HS-20094 Injection — HS-20094 injected subcutaneously once weekly
  Arms: Treatment Group A; Treatment Group B
Drug: Dulaglutide Injection — Dulaglutide injected subcutaneously once weekly
  Arms: Treatment Group C

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of HS-20094 once weekly (QW) in subjects with type 2 diabetes mellitus not adequately controlled with metformin monotherapy or in combination with SGLT2 inhibitors compared to Dulaglutide QW for 44 weeks and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, Age ≥18 years at the time of signing informed consent.
2. Stable daily dose(s) for ≥90 days prior to screening of : 1) Any metformin formulations ≥1500 mg daily or maximum tolerated (≥1000mg daily). 2) Any metformin formulations ≥1500 mg daily or maximum tolerated (≥1000mg daily) with one type of SGLT-2 inhibitors;
3. Glycated hemoglobin was 7.5% ≤HbA1c ≤11.0%;
4. BMI ≥ 23 kg/m2.

Exclusion Criteria:

1. Uncontrollable hypertension(with or without antihypertensive treatment) : systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg at screening.
2. Diagnosed or suspected with type 1 diabetes mellitus, special types of diabetes or secondary diabetes.
3. History of significant hematological disorders (e.g., sickle cell disease, hemolytic anemia, myelodysplastic syndrome, etc.) or other conditions causing hemolysis or instability of red blood cells (e.g., malaria, hypersplenism, etc.).
4. Presence of an endocrine disorder or history that may significantly affect bady weight(e.g., Cushing's syndrome, hypothyroidism or hyperthyroidism, except hypothyroidism if thyroid hormone replacement dose has been stable for at least 6 months) ；
5. Severe infection, severe trauma, or moderate-to-major surgery within 4 weeks before screening.
6. Participated in clinical trials of any drug or medical device within 12 weeks prior to screening, and participation in clinical trials is defined as signing informed consent and using investigational drugs (including placebo) or investigational medical devices; Or is still in the trial drug within 5 half-lives (whichever is Longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Week 0 to Week 44
  Change from baseline in HbA1c after 44 weeks of treatment

SECONDARY OUTCOMES:
Proportion of subjects with HbA1c<7.0% and ≤6.5% | Week 0 to Week 44
  Proportion of subjects with HbA1c<7.0% and ≤6.5% after 44 weeks of treatment
Change in FPG | Week 0 to Week 44
  Change from baseline in FPG after 44 weeks of treatment
Change in body weight | Week 0 to Week 44
  Change from baseline in Change in body weight after 44 weeks of treatment
Proportion of subjects with weight loss ≥5% and ≥10% | Week 0 to Week 44.
  Proportion of subjects with weight loss ≥5% and ≥10% after 44 weeks of treatment
Change in HbA1c | Week 0 to Week 52
  Change from baseline in HbA1c after 52 weeks of treatment
Proportion of subjects with HbA1c<7.0% and ≤6.5% | Week 0 to Week 52
  Proportion of subjects with HbA1c<7.0% and ≤6.5% after 52 weeks of treatment
Change in FPG | Week 0 to Week 52
  Change from baseline in FPG after 52 weeks of treatment
Change in body weight | Week 0 to Week 52
  Change from baseline in Change in body weight after 52 weeks of treatment
Proportion of subjects with weight loss ≥5% and ≥10% | Week 0 to Week 52
  Proportion of subjects with weight loss ≥5% and ≥10% after 52 weeks of treatment
Incidence and severity of adverse events | Week 0 to Week 52+4 weeks follow-up
  Severity (mild, moderate and severe) is assessed by investigator

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shandong Provincial Hospital, Jinan, Shandong
  - Tianjin Medical University General Hospital (Zhu Xianyi Memorial Hospital), Tianjin, Tianjn